CLINICAL TRIAL: NCT04631341
Title: The Intervention Effect Of Melatonin On The Risk Of Cardiovascular Events And Malignant Tumors In The Elderly: A Prospective, Randomized Parallel Controlled Study Based On Large Cohorts
Brief Title: Melatonin and Risk Of Cardiovascular Events And Malignant Tumors In The Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tongji Hospital (Other); Huadong Hospital (Other); ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Jun Pu, Director of Cardiovascular Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Melatonin Intervention Study
Record Dates: First submitted 2020-08-16; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases
Keywords: Cohort study; Natural Population; China
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin Group (Experimental): Take melatonin supplements
  Interventions: Dietary Supplement: Melatonin
- Normal Control Group (No Intervention): Don't take melatonin supplements

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin 5mg every night, for one year
  Arms: Melatonin Group

SUMMARY:
Cardiovascular diseases and tumors seriously threaten human health. There are many risk factors that affect the occurrence and death of cardiovascular diseases and malignant tumors. In addition to genetic and congenital factors, it also includes bad lifestyles, such as smoking, drinking, abnormal metabolism, excessive stress, etc. Many factors such as excessive stress and staying up late can cause abnormal circadian rhythms. The regulation of circadian rhythm is likely to be a key key to the early prevention of cardiovascular diseases and tumors.

Melatonin has an important role in regulating the circadian rhythm of the human body. The latest research of our research group confirmed that melatonin can reduce the level of oxidative stress through the retinoic acid-related orphan nuclear receptor alpha (RORα) and thereby inhibit pathological cardiac hypertrophy; melatonin can regulate the polarization and polarization of macrophages RORα receptor stabilizes vulnerable plaque in arteries and prevents plaque rupture.

In China, melatonin is widely used in the market as a health product. However, the protective mechanism of melatonin in cardiovascular diseases and tumors is still unclear, and large-scale population intervention studies are still lacking. The level of melatonin in the daytime changes little with age, but the peak at night gradually decreases with age. In people aged 60 and above, the peak of melatonin at night decreased significantly. We speculate that melatonin supplementation may be able to reduce the oxidative damage of mitochondria by maintaining the level of melatonin at night in the body, delay cell decay, and delay this physiological process.

Therefore, the project team intends to combine the developed new cardiovascular disease and tumor risk prediction models in the Shanghai elderly cohort established in the early stage, and randomize groups of healthy people in the same risk stratification, according to whether or not to supplement melatonin. There are two cohorts: the melatonin intervention cohort and the parallel control cohort. By observing the efficacy indicators of cardiovascular disease and tumor incidence in the two groups during the follow-up period, it provides evidence-based medical evidence for the future clinical application of melatonin.

DETAILED DESCRIPTION:
Cardiovascular diseases and tumors seriously threaten human health. With the aging of the population in my country, the number of patients with two diseases has been increasing year by year, the difficulty of treatment has greatly increased, and the prognosis of most patients is poor. Therefore, it is of great clinical significance to explore safe and effective intervention programs to prevent cardiovascular diseases and malignant tumors in the elderly.

There are many risk factors that affect the occurrence and death of cardiovascular diseases and malignant tumors. In addition to genetic and congenital factors, it also includes bad lifestyles, such as smoking, drinking, abnormal metabolism, excessive stress, etc. Many factors such as excessive stress and staying up late can cause abnormal circadian rhythms [5, 6]. The regulation of circadian rhythm is likely to be a key key to the early prevention of cardiovascular diseases and tumors.

Melatonin has an important role in regulating the circadian rhythm of the human body. A number of basic and clinical studies at home and abroad have shown that melatonin has a protective effect on inhibiting cardiovascular disease and tumor occurrence. The latest research of our research group confirmed that melatonin can reduce the level of oxidative stress through the retinoic acid-related orphan nuclear receptor alpha (RORα) and thereby inhibit pathological cardiac hypertrophy; melatonin can regulate the polarization and polarization of macrophages RORα receptor stabilizes vulnerable plaque in arteries and prevents plaque rupture.

In China, melatonin is widely used in the market as a health product. Melatonin has a wide range of sources, no obvious toxic and side effects to the body, and high bioavailability, which suggests that it can prevent cardiovascular diseases and It has important potential in the occurrence of tumors. However, the protective mechanism of melatonin in cardiovascular diseases and tumors is still unclear, and large-scale population intervention studies are still lacking. The level of melatonin in the daytime changes little with age, but the peak at night gradually decreases with age. In people aged 60 and above, the peak of melatonin at night decreased significantly. We speculate that melatonin supplementation may be able to reduce the oxidative damage of mitochondria by maintaining the level of melatonin at night in the body, delay cell decay, and delay this physiological process.

Therefore, the project team intends to combine the developed new cardiovascular disease and tumor risk prediction models in the Shanghai elderly cohort established in the early stage, and randomize groups of healthy people in the same risk stratification, according to whether or not to supplement melatonin. There are two cohorts: the melatonin intervention cohort and the parallel control cohort. By observing the efficacy indicators of cardiovascular disease and tumor incidence in the two groups during the follow-up period, it provides evidence-based medical evidence for the future clinical application of melatonin.

ELIGIBILITY:
Inclusion Criteria:

1. Queue members;
2. Han nationality;
3. Between 60-74 years old, no gender limit;
4. Women are in menopause;
5. Patients without a history of malignant tumors (except for non-melanoma skin cancer), myocardial infarction, stroke, transient ischemic attack (TIA), angina, coronary artery bypass graft (CABG) or Percutaneous Coronary Intervention;
6. No mental illness;
7. No history of supplement allergy or supplement allergy;
8. Subjects voluntarily participate in this study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. People who have difficulty swallowing or have known supplementary malabsorption;
2. Have received any other clinical trial treatment within 1 year;
3. The subject has a known, active or suspicious autoimmune disease;
4. The subject has severe infections, including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.;
5. The subject has used a live attenuated vaccine in the past 30 days;
6. The subject has been taking antidepressant medication before or is taking;
7. Use of anticoagulants at baseline, history of kidney stones, renal failure or dialysis, hypercalcemia, hypoparathyroidism or hyperthyroidism, severe liver disease (cirrhosis), sarcoidosis or other granulomatous diseases, such as Active chronic tuberculosis or Wegener's granulomatosis, dementia, epilepsy, rheumatoid arthritis, sleep apnea syndrome, alcoholism;
8. Situations deemed unsuitable by other researchers.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total cancer and cardiovascular disease incidence | up to five years
  The primary cancer endpoint will be total cancer incidence (excluding non-melanoma skin cancer). For cardiovascular disease (CVD), the primary endpoint will be a composite endpoint of myocardial infarction, stroke, and CVD incidence.

SECONDARY OUTCOMES:
Cancer mortality and a composite endpoint adding revascularization procedures of coronary artery bypass grafting and percutaneous coronary intervention | up to five years
  Secondary endpoints will include cancer mortality and the individual sites of colorectal, breast, and prostate cancer.
  A second composite endpoint adding revascularization procedures of coronary artery bypass grafting and percutaneous coronary intervention, as well as the individual endpoints of myocardial infarction, stroke, revascularization, and CVD mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD,PhD, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu L, Su Y, Zhao Y, Sheng X, Tong R, Ying X, Gao L, Ji Q, Gao Y, Yan Y, Yuan A, Wu F, Lan F, Pu J. Melatonin differentially regulates pathological and physiological cardiac hypertrophy: Crucial role of circadian nuclear receptor RORalpha signaling. J Pineal Res. 2019 Sep;67(2):e12579. doi: 10.1111/jpi.12579. Epub 2019 Apr 24. PMID 30958896
- [Background] Ding S, Lin N, Sheng X, Zhao Y, Su Y, Xu L, Tong R, Yan Y, Fu Y, He J, Gao Y, Yuan A, Ye L, Reiter RJ, Pu J. Melatonin stabilizes rupture-prone vulnerable plaques via regulating macrophage polarization in a nuclear circadian receptor RORalpha-dependent manner. J Pineal Res. 2019 Sep;67(2):e12581. doi: 10.1111/jpi.12581. Epub 2019 May 14. PMID 31009101
- [Background] Zhao Y, Xu L, Ding S, Lin N, Ji Q, Gao L, Su Y, He B, Pu J. Novel protective role of the circadian nuclear receptor retinoic acid-related orphan receptor-alpha in diabetic cardiomyopathy. J Pineal Res. 2017 Apr;62(3). doi: 10.1111/jpi.12378. Epub 2017 Feb 22. PMID 27862268
- [Background] Zhao YC, Xu LW, Ding S, Ji QQ, Lin N, He Q, Gao LC, Su YY, Pu J, He B. Nuclear receptor retinoid-related orphan receptor alpha deficiency exacerbates high-fat diet-induced cardiac dysfunction despite improving metabolic abnormality. Biochim Biophys Acta Mol Basis Dis. 2017 Aug;1863(8):1991-2000. doi: 10.1016/j.bbadis.2016.10.029. Epub 2016 Nov 5. PMID 27825849
- [Background] He B, Zhao Y, Xu L, Gao L, Su Y, Lin N, Pu J. The nuclear melatonin receptor RORalpha is a novel endogenous defender against myocardial ischemia/reperfusion injury. J Pineal Res. 2016 Apr;60(3):313-26. doi: 10.1111/jpi.12312. Epub 2016 Feb 16. PMID 26797926